CLINICAL TRIAL: NCT00984698
Title: A Trial of Group Psychotherapy for Veterans and Military Personnel With Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Southern Arizona VA Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tricia Haynes, Assistant Professor, Dept of Psychiatry, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH-08-2-0121
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-02

CONDITIONS: Posttraumatic Stress Disorder; Depression; Insomnia Disorder
Keywords: Posttraumatic Stress Disorder; Depression; Sleep Initiation and Maintenance Disorders; Insomnia; Psychotherapy, Group; Cognitive Behavioral Therapy; Randomized Controlled Trial; Veterans; Social Rhythms
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Structured Therapy (Experimental): Cognitive Behavioral Social Rhythm Group Therapy is designed to improve mood and sleep by stabilizing social rhythms, increasing exposure to ambient light, changing dysfunctional bed/bedtime associations, activating the imagery system by changing nightmare content, and challenging dysfunctional automatic thoughts that might contribute to behavioral inactivation and nonadherence to the therapy protocol. There is no discussion of past traumatic events.
  Interventions: Behavioral: Cognitive Behavioral Social Rhythm Group Therapy
- Unstructured Therapy (Active Comparator): Present Centered Group Therapy includes education about the typical symptoms and features associated with PTSD and MDD, with a focus on how these symptoms affect interpersonal relationships. It uses the group format to decrease isolation, normalize symptoms, and provide the experience of giving and receiving support. Some relaxation training is provided early in therapy. There is no discussion of past traumatic events.
  Interventions: Behavioral: Present Centered Group Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Social Rhythm Group Therapy — 12 weeks, 2h structured group therapy
  Arms: Structured Therapy
Behavioral: Present Centered Group Therapy — 12 weeks, 2h relatively unstructured group therapy
  Arms: Unstructured Therapy

SUMMARY:
The purpose of this study is to test the effectiveness of group psychotherapy designed specifically for male veterans and active-duty personnel with Post-traumatic Stress Disorder (PTSD), Major Depressive Disorder (MDD) and with disturbances in their sleep or daily routine.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness of a group psychotherapy designed specifically for male veterans and active-duty personnel with Post-traumatic Stress Disorder (PTSD), Major Depressive Disorder (MDD) and with disturbances in their sleep or daily routine. We will compare two group therapies, one of which has been examined in previous studies for veterans with PTSD. Both group therapies have been shown to reduce symptoms of anxiety and depression in some veterans. However, neither group therapy has been proven to be more effective than treatment as usual for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Veteran or active duty military personnel
* Current posttraumatic stress disorder (PTSD), at least moderate severity
* Criterion A exposure to trauma occurring after the age of 18
* Major depressive disorder (MDD), at least moderate severity
* Disturbances in sleep (primary insomnia, insomnia related to PTSD, or nightmare disorder) or daily routine

Exclusion Criteria:

* Current or past bipolar disorder
* Current psychotic disorder
* Substance abuse/dependence in last 30 days
* Uncontrolled serious medical condition or neurological disorder
* Currently working an overnight shift
* Primary untreated sleep apnea, restless legs syndrome

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Haynes, PhD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Southern Arizona VA Healthcare System (SAVAHCS), Tucson, Arizona
  - University of Arizona, Tucson, Arizona

REFERENCES:
- [Derived] Haynes PL, Burger SB, Kelly M, Emert S, Perkins S, Shea MT. Cognitive behavioral social rhythm group therapy versus present centered group therapy for veterans with posttraumatic stress disorder and major depressive disorder: A randomized controlled pilot trial. J Affect Disord. 2020 Dec 1;277:800-809. doi: 10.1016/j.jad.2020.09.009. Epub 2020 Sep 7. PMID 33065820

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans were recruited from the Southern Arizona VA Health Care System, Mental Health Clinic, September 2009 to July 2011.
Pre-assignment Details: 115 enrolled, 50 eligible, 7 withdrew prior to randomization (3 time commitment, 2 lost contact, 1 changed mind/unknown, 1 travel distance)
Groups:
- Cognitive Behavioral Social Rhythm Group Therapy: CBSRT is designed to improve mood and sleep by stabilizing social rhythms, increasing exposure to ambient light, changing dysfunctional bed/bedtime associations, activating the imagery system by changing nightmare content, and challenging dysfunctional automatic thoughts that might contribute to behavioral inactivation and nonadherence to the therapy protocol. There is no discussion of past traumatic events.
- Present Centered Group Therapy: PCGT includes education about the typical symptoms and features associated with PTSD and MDD, with a focus on how these symptoms affect interpersonal relationships. It uses the group format to decrease isolation, normalize symptoms, and provide the experience of giving and receiving support. Some relaxation training is provided early in therapy. There is no discussion of past traumatic events.
Period: Overall Study
Arm/Group | Cognitive Behavioral Social Rhythm Group Therapy | Present Centered Group Therapy
Started | 21 | 22
Completed | 18 | 14
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Social Rhythm Group Therapy | Present Centered Group Therapy | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 22 | 43
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.24 (13.99) | 51.46 (12.60) | 48.42 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 22 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Secondary Outcome: PTSD
Description: Clinician-Administered PTSD Scale (CAPS), DSM-IV The CAPS is a 17-item interview assessment post-traumatic stress disorder (PTSD) symptom severity. Total score ranges from 0 (no PTSD symptoms) to 136 (maximum PTSD symptoms).
Time Frame: post-treatment, at 12 weeks
Population: CBSRT arm: 18 participants who completed 75% of psychotherapy sessions; 20 participants who completed 12-week post-treatment assessment
  PCGT arm: 14 participants who completed 75% of psychotherapy sessions; 17 participants who completed 12-week post-treatment assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Social Rhythm Group Therapy | Present Centered Group Therapy
Number analyzed (Participants) | 20 | 17
units on a scale | 67.35 (26.82) | 62.47 (24.83)
Statistical Analysis 1: Comparison: Cognitive Behavioral Social Rhythm Group Therapy vs Present Centered Group Therapy; Analysis must be qualified by small sample size, worse baseline symptom severity in CBSRT arm, and greater levels of attrition in PCGT arm; Test type: Superiority or Other; p < .05, Mixed Models Analysis

2. Primary Outcome: Depression
Description: Hamilton Rating Scale for Depression, 17 item The Hamilton Rating Scale for Depression is an interview assessment of depression symptom severity. Total score range is from 0 (no symptoms of depression) to 52 (maximum symptoms of depression).
Time Frame: post-treatment, at 12 weeks
Population: CBSRT arm: 18 participants completed 75% of psychotherapy sessions; 20 participants completed study assessment at 12-week post-treatment time point
  PCGT arm: 14 participants completed 75% of psychotherapy sessions; 17 participants completed study assessment at 12-week post-treatment time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Social Rhythm Group Therapy | Present Centered Group Therapy
Number analyzed (Participants) | 20 | 17
units on a scale | 20.30 (6.51) | 19.18 (5.79)
Statistical Analysis 1: Comparison: Cognitive Behavioral Social Rhythm Group Therapy vs Present Centered Group Therapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .05, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Cognitive Behavioral Social Rhythm Group Therapy | Present Centered Group Therapy
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes